CLINICAL TRIAL: NCT07216651
Title: WeDosify Real-World Evidence: Evaluating a Clinical Decision Support and Patient Engagement Tool for Personalized Semaglutide Dosing in Adults With Overweight or Obesity in the United States
Brief Title: WeDosify Real World Evidence (RWE) Study: Personalized Semaglutide Dosing in U.S. Adults
Status: Recruiting | Type: Observational
Sponsor: Closed Loop Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: CLM-OB-001
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obesity & Overweight
Keywords: Obesity; Overweight; GLP-1; Semaglutide
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational semaglutide treated cohort: This research focuses on adult subjects who have recently been prescribed semaglutide (Wegovy) for obesity or overweight.

SUMMARY:
This research study is studying WeDosify, an interactive web-based Clinical Decision Support tool that assists healthcare professionals in managing adults with excess weight or obesity using a Glucagon-like peptide-1 (GLP-1) drug treatment such as semaglutide.

DETAILED DESCRIPTION:
Researchers at Amarillo Premier Research, working with Closed Loop Medicine Ltd (CLM), want to improve how excess weight and obesity are managed. There is a need for tools that support more consistent, data-informed and personalized treatment decisions in weight management. This research focuses on subjects who have recently been prescribed semaglutide (Wegovy). Semaglutide is a widely used medicine that helps patients to lose excess weight and belongs to a group of medicines called Glucagon-like peptide 1s (GLP-1s).

Only subjects who are receiving semaglutide treatment as part of their routine weight management will be invited by the study doctor to join this research study. Once consented, the study doctor will have access to a product called WeDosify, an interactive web-based Clinical Decision Support tool that assists healthcare professionals in managing adults with excess weight or obesity using GLP-1 treatment.

Participation in this study will last approximately 3 months and will include approximately 4 consultations, either study visits to the research center or remote consultations

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older.
2. Participants must have a diagnosis of either obesity or overweight.
3. Participants must have initiated first-time semaglutide treatment within the past 4-12 weeks for the management of overweight or obesity, in line with United States Prescribing Information (USPI) and the clinical judgment of the responsible Healthcare Professional (HCP).
4. Participants must have access to and be able to use suitable weighing scales to record their weight before or during consultations.
5. Participants must provide written informed consent to participate in this study, including agreeing to adhere to the associated procedures.

Exclusion Criteria:

1. Participants with conditions that the Healthcare Professional (HCP) deems would prevent effective use of weighing scales and accurate self-monitoring or reporting of body weight.
2. Failure to satisfy the responsible Healthcare Professional (HCP) of fitness to participate for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Obesity or Overweight receiving semaglutide (Wegovy)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who persisted on semaglutide treatment over the study period | 3 months
  The primary outcome is treatment persistence during the 3-month observation period, defined as the proportion of participants who remain on semaglutide treatment without discontinuation. Discontinuation will be defined as either a formal cessation of medication or the absence of a prescription renewal within the expected timeframe

SECONDARY OUTCOMES:
Number and percentage of participants discontinuing semaglutide due to unwanted side effects or other clinically significant reasons | 3 months
  Number and percentage of participants discontinuing semaglutide due to unwanted side effects or other clinically significant reasons measured as number and proportion of participants stopping semaglutide and the documented reason for discontinuation
Weight loss from baseline to end of study | 3 months
  Weight loss from baseline to end of study comprising weight loss magnitude and rate, assessed by absolute and percentage change in body weight
Patients' experience of WeDosify and perceived impact of treatment using custom Patient-Reported Experience Measure (PREM) and Patient-Reported Outcome Measure (PROM) questionnaires at end of study | 3 months
  At the end of the study, participants will complete a brief e-questionnaire to capture their experience of the WeDosify-supported treatment journey.
  The questionnaire will use 5-point Likert scale and free text questions to assess:
  * Patient-Reported Outcome Measures (PROMs): to assess the perceived impact of WeDosify on weight and overall health.
  * Patient-Reported Experience Measures (PREMs): to capture satisfaction with WeDosify, including engagement with treatment, clarity of the treatment plan, and motivation to complete it.
Healthcare Professional (HCP) user experience and perceived utility assessed by custom questionnaire at end of study (to include utilization and ease of use) | 3 months
  The Healthcare Professional (HCP) will complete a custom e-questionnaire at the end of the study to capture their overall experience of using the WeDosify tool.
  This e-questionnaire will use 5-point Likert scale and free text questions to assess:
  * Usability and ease of use
  * Perceived value of the treatment options
  * HCP insights on clinical use and potential improvements

CONTACTS AND LOCATIONS:
Overall Officials: Susan Neese, MD, Principal Investigator — Amarillo Premier Research
Locations (1):
- Amarillo Premier Research (an Objective Health Partnership), Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided